CLINICAL TRIAL: NCT01535625
Title: Clinical Evaluation of the Momo Cobalt-Chromium Coronary Stent System for the Treatment of Patients With Coronary Artery Disease
Brief Title: Safety and Effectiveness of the Coronary Momo Stent
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: be Medical (Industry)
Collaborators: Japan Stent Technology Europe GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BM-MOMO-04-001
Record Dates: First submitted 2012-02-15; First posted 2012-02-20 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Atherosclerosis; CAD
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Momo stent (Other): Patients with PCI
  Interventions: Device: Momo stent

INTERVENTIONS:
Device: Momo stent — Patients with PCI

SUMMARY:
This study evaluates the safety and effectiveness of the Momo Cobalt Chromium stent system for the treatment of single de novo lesions in a native coronary artery. The stent is coated with diamond-like carbon to decrease the risk of acute and late stent thrombosis, to increase the resistance towards corrosion and to significantly improve endothelialisation through the inhibition of elution of metallic ions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stable angina pectoris (Canadian Cardiovascular Society [CCS] I to IV) or unstable angina pectoris (Braunwald classification IB-C, IIB-C or IIIB-C) or patients with documented silent ischemia.
2. Patients who are eligible for coronary revascularization by angioplasty and stenting and by CABG (if required as bail-out).
3. Patients with a de novo lesion in a native coronary artery between > 50 % and < 100 % stenosis.
4. One or two heart vessel disease with a maximum of 2 lesions to be treated by stenting.

   Both lesions have to be treated with study stents.
5. Target vessel suitable for implantation of a single stent with a target vessel diameter of ≥ 2.5 mm and lesion length < 20 mm.
6. Patients with left ventricular ejection fraction (LVEF) of > 30 %.
7. Patients willing to sign a written informed consent prior to participation and willing to be compliant with all requested follow-up evaluations.

Exclusion Criteria:

1. Patients under the age of 18 or unable to give informed consent.
2. Women of child bearing potential.
3. Patients who currently participate in another study (whatever the subject of that study is).
4. Patients who participated in another investigational cardiovascular drug or device study, which have not completed the primary endpoint follow-up period within the past 30 days.
5. Patients with a life expectancy of less than 24 months or factors making clinical and/or angiographic follow-up difficult (no fixed address, etc.).
6. Patients who intend to have a major (as per principal investigators' medical judgment) surgical intervention within 6 months of enrolment in the study.
7. Patients with an episode of sustained ischemic chest pain exceeding 15 minutes duration within 24 hours prior to stenting or patients with new ST elevation within 48 hours prior to stenting.
8. Patients with a contraindication to emergency coronary bypass surgery.
9. Any individual who may refuse a blood transfusion.
10. Patients with serum creatinine > 2.0 mg/dl or (> 180 µmol/l).
11. Patients with a baseline platelet count less than 100,000 platelets/mm³.
12. Patients with intolerance or contraindication to acetylsalicylic acid (aspirin), heparin, clopidogrel or ticlopidine drug therapy.
13. Patients with contrast agent hypersensitivity that cannot be adequately pre-medicated.
14. Patients whose target vessel has been stented before.
15. Any procedure to treat another coronary artery scheduled within 6 months after implantation of the study stent.

Exclusion criteria related to angiography

1. Patients with previous PCI of the same segment (i.e. no restenotic lesions).
2. Any previous interventional procedure (less than 6 months) anywhere within the target vessel.
3. Target lesion is located in or supplied by an arterial or venous bypass graft
4. Target lesion involves a side branch ≥ 2.0 mm in diameter.
5. Ostial target lesion (within 3.0 mm of vessel origin).
6. Target vessel has evidence of thrombus or is excessively tortuous that makes it unsuitable for proper stent delivery and deployment.
7. Patients with total occlusions (TIMI 0).
8. Significant (>50%) stenosis proximal or distal to the target lesion than might require revascularization or impede run off.
9. Target lesion requires treatment with a device other than the predilatation balloon prior to stent placement (including but not limited to, directional coronary atherectomy, excimer laser, rotational atherectomy, cutting balloon etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-01 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
6-month angiography | 6 months
  Binary restenosis(defined as >50% diameter stenosis by QCA), late loss, percent diameter stenosis, minimal lumen diameter

SECONDARY OUTCOMES:
Major adverse cardiac events | 6 months
  including death, recurrent non-fatal myocardial infarction, emergent CABG and/or clinically driven target vessel revascularization
MACE | 1 month, 6 months, 12 months
  Including death, recurrent non-fatal myocardial infarction, emergent CABG and/or clinically driven target vessel revascularization, target lesion revascularization (TLR), target vessel revascularization (TVR), target vessel failure (TVF) and stent thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Luc Janssens, MD, Principal Investigator — Imelda vzw
Locations (6):
- Belgium (6):
  - ZNA Middelheim, Antwerp
  - Imelda vzw, Bonheiden
  - AZ Sint Jan, Bruges
  - UZ Brussel, Brussels
  - Ziekenhuis Oost-Limburg, Genk
  - AZ Maria Middelares, Ghent